CLINICAL TRIAL: NCT05605860
Title: Development of a Predictive Algorithm for a Hemoglobin Value of Less Than 10 g/dl Postoperatively in Scheduled Hip or Knee Arthroplasty
Acronym: Predi_Hb
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Predi_Hb
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-02

CONDITIONS: Hip Prosthetic Surgery; Knee Prosthetic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hip (THR) or knee (KT) prosthetic surgery is a bleeding surgery with an average blood spoliation of about 1 liter and an average decrease of about 3 g/dl in hemoglobinemia (Hb). Consequently, anemia is observed postoperatively in almost all patients (between 85% and 99% depending on the preoperative Hb value). In all cases, anemia-related events delay the patient's recovery, favor the occurrence of complications and prolong the length of stay. The immediate treatment of acute postoperative anemia is based on transfusion of red blood cells (RBCs). However, this presents several risks for the patient. The first is immediate and associated with the procedure: risk of error with ABO/Rhesus incompatibility, sepsis, pulmonary edema, etc. The second is a medium-term risk, with an increased risk of infection after prosthetic hip or knee surgery. In the long term, immediate postoperative blood transfusion is associated with higher mortality. In order to reduce the likelihood of a patient receiving RGCs, strategies have been developed within a "Patient Blood Management" (PBM), which could be translated as "Personalized Blood Transfusion Management". This strategy is based on 3 pillars: preoperatively, to ensure a patient's hemoglobin level of at least 13 g/dl; during the procedure, to limit blood loss; and postoperatively, to limit the indications for blood transfusion and the number of RGCs to the strict necessary. As the main determinant to trigger the prescription of a blood transfusion is the Hb value, the objective is that the lowest value of hemoglobinemia (Hb_nadir) postoperatively is as close as possible to 10 g/dl. The objective of this study is to describe, by means of the data available in the computerized patient record of patients undergoing scheduled THR or PTG operations at the Paris Saint Joseph Hospital, a prediction equation for Hb_nadir < 10 g/dl and, thus, to prescribe iron and ESAs only in patients who require them.

ELIGIBILITY:
Inclusion Criteria:

- Patient operated on for elective hip or knee arthroplasty within the Paris Saint Joseph hospital site (HPSJ) between January 1, 2019 and December 31, 2021. Over the 36-month period, 1281 patients underwent THP (approximately 60%) or TKP (approximately 40%) surgery.

Exclusion Criteria:

* Patient who received iron infusion and/or injections of erythropoiesis stimulating agents within one month prior to surgery
* Patient who received an infusion of packed red blood cells in the month prior to surgery
* Absence of preoperative hemoglobinemia
* No postoperative hemoglobinemia
* Patient who had surgery in the previous month
* Patient operated on both sides (hip or knee) during the same operation
* Patient operated in emergency
* Patient with a hereditary anemia
* Patient opposing the use of his data for this research
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patient operated on for elective hip or knee arthroplasty within the Paris Saint Joseph hospital site (HPSJ) between January 1, 2019 and December 31, 2021. Over the 36-month period, 1281 patients underwent THP (approximately 60%) or TKP (approximately 40%) surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1041 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Validation of the statistical model for predicting patients with a postoperative hemoglobin value (Hb_nadir) will be < 10 g/dl | Year1
  This outcome corresponds to the Quality of the prediction obtained on the validation cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal ALFONSI, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Spahn DR. Anemia and patient blood management in hip and knee surgery: a systematic review of the literature. Anesthesiology. 2010 Aug;113(2):482-95. doi: 10.1097/ALN.0b013e3181e08e97. PMID 20613475
- [Background] Lasocki S, Krauspe R, von Heymann C, Mezzacasa A, Chainey S, Spahn DR. PREPARE: the prevalence of perioperative anaemia and need for patient blood management in elective orthopaedic surgery: a multicentre, observational study. Eur J Anaesthesiol. 2015 Mar;32(3):160-7. doi: 10.1097/EJA.0000000000000202. PMID 25564780
- [Background] Kim JL, Park JH, Han SB, Cho IY, Jang KM. Allogeneic Blood Transfusion Is a Significant Risk Factor for Surgical-Site Infection Following Total Hip and Knee Arthroplasty: A Meta-Analysis. J Arthroplasty. 2017 Jan;32(1):320-325. doi: 10.1016/j.arth.2016.08.026. Epub 2016 Aug 31. PMID 27682006
- [Background] Smilowitz NR, Oberweis BS, Nukala S, Rosenberg A, Zhao S, Xu J, Stuchin S, Iorio R, Errico T, Radford MJ, Berger JS. Association Between Anemia, Bleeding, and Transfusion with Long-term Mortality Following Noncardiac Surgery. Am J Med. 2016 Mar;129(3):315-23.e2. doi: 10.1016/j.amjmed.2015.10.012. Epub 2015 Oct 30. PMID 26524702
- [Background] Roque-Castellano C, Marchena-Gomez J, Farina-Castro R, Acosta-Merida MA, Armas-Ojeda MD, Sanchez-Guedez MI. Perioperative Blood Transfusion is Associated with an Increased Mortality in Older Surgical Patients. World J Surg. 2016 Aug;40(8):1795-801. doi: 10.1007/s00268-016-3521-2. PMID 27142623
- [Background] Jans O, Jorgensen C, Kehlet H, Johansson PI; Lundbeck Foundation Centre for Fast-track Hip and Knee Replacement Collaborative Group. Role of preoperative anemia for risk of transfusion and postoperative morbidity in fast-track hip and knee arthroplasty. Transfusion. 2014 Mar;54(3):717-26. doi: 10.1111/trf.12332. Epub 2013 Jul 5. PMID 23829298